CLINICAL TRIAL: NCT04858659
Title: A Multi-center, Randomized, Double-blind, Active-controlled, Parallel-designed, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of PK101 Compared With PK101-002 in Patients With Knee Osteoarthritis
Brief Title: A Phase 3 Study to Assess the Efficacy and Safety of PK101 in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PMG Pharm Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PK101_P301
Record Dates: First submitted 2021-04-05; First posted 2021-04-26 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PK101 group (Experimental)
  Interventions: Drug: PK101; Drug: PK101-002 placebo
- PK101-002 group (Active Comparator)
  Interventions: Drug: PK101-002; Drug: PK101 placebo

INTERVENTIONS:
Drug: PK101 — 1 tablet at each time, 2 times a day
  Arms: PK101 group
Drug: PK101-002 — 1 tablet at each time, 2 times a day
  Arms: PK101-002 group
Drug: PK101 placebo — 1 tablet at each time, 2 times a day
  Arms: PK101-002 group
Drug: PK101-002 placebo — 1 tablet at each time, 2 times a day
  Arms: PK101 group

SUMMARY:
The purpose of this study is to compare the efficacy and the safety of PK101 in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the efficacy of PK101 compared with PK101-002 at Week 8 in osteoarthritis. Also evaluates the safety of PK101.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥40 and of age
* Patients who meets the American College Rheumatology (ACR) criteria and has lasted for at least three months after diagnosis of one-sided or bilateral knee osteoarthritis.
* Radiographic evidence of grade 1 ~ 3 osteoarthritis based on the Kellgren & Lawrence radiographic entry criteria at visit 1
* Score of 100mm pain VAS ≤ 80mm at visit 1
* Written consent form voluntarily
* Score of 100mm pain VAS ≥ 40mm at visit 3
* Patients with an individual medication compliance of 70% or more of the IP administered during the Run-in period

Exclusion Criteria:

* Patients who has a history of hypersensitivity to components of IP, NSAIDs including COX-2 inhibitors, a history of hypersensitivity to aspirin, or allergic reactions to sulfonamides
* Patients with inflammatory, infectious, metabolic, septic arthritis or rheumatoid arthritis other than osteoarthritis
* Patients with a condition that can affect the joints
* Patients who have undergone arthroscopic surgery within 1 year , knee joint surgery within 5 years, synoviorthesis within 3 months prior to visit 1 to the target knee, or who have planned surgery during the trial period
* Patients who have used corticosteroids as follows:

  * Inj. of corticosteroid, including intraarticular administration, into the target knee within 3 months prior to visit 1
  * Oral corticosteroid administration within 1 month prior to visit 1
* Patients who have intraarticular injected hyaluronic acid or cell therapy products, gene therapy products, etc. for the treatment of osteoarthritis within 3 months prior to visit 1

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Change during activity in 100mm Pain VAS | baseline through week 8
  Visual Analogue Scale, 0 mm no pain, 100 mm worst pain ever

SECONDARY OUTCOMES:
Change during activity in 100mm Pain VAS | baseline through week 4
  Visual Analogue Scale, 0 mm no pain, 100 mm worst pain ever
Change at rest in 100mm Pain VAS | baseline through week 4, 8
  Visual Analogue Scale, 0 mm no pain, 100 mm worst pain ever
Change in WOMAC(Western Ontario and McMaster Universities Osteoarthritis Index using the Visual Analogue Scale, Version 3.1) sub scale & total score | baseline through week 4, 8
  Assessment of pain, stiffness and physical function. Score range 0-500 mm for Pain, 0-200 mm for Stiffness, and 0-1700 mm for Physical Function. Higher scores indicate worse pain, stiffness, and functional limitations.
Change in PGA | baseline through week 8
  PGA for disease severity (Patient's Global Assessment, 1=Very good, 2=Good, 3=Fair, 4=Poor, 5=Very Poor)
Change in SF-36 sub scale & PCS, MCS as measured by Health Survey(Short Form, SF-36 v2, Physical Component Summary, Mental Component Summary) | baseline through week 8
  The SF-36 v2 is a 36-item, patient-reported survey of patient's health, consisting of 2 components(the PCS and the MCS) included 8 subscales.
  Patients rated their QoL using a 2-6 point Likert Scale. Score is converting the original score to 0~100 points.
  The lower score means poor health status, and the higher score, the better.

CONTACTS AND LOCATIONS:
Locations (1):
- Jeonbuk National University Hospital, Jeonju, South Korea